CLINICAL TRIAL: NCT05277233
Title: Endothelial Dysfunction and Cardiovascular Risk After Preeclampsia
Brief Title: Cardiovascular Risk After Preeclampsia
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Kristin Kraeker, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: CARPE
Record Dates: First submitted 2022-02-18; First posted 2022-03-14 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Plasma, serum, peripheral blood mononuclear cells (PBMCs)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Early-onset preeclampsia: Defined as preeclampsia that develops before 34 weeks of gestation
- Late-onset preeclampsia: Defined as preeclampsia that develops after 34 weeks of gestation
- Control: Healthy pregnancies, matched to early and late-onset cases

SUMMARY:
Investigation of cardiovascular risk 5-15 years after early or late-onset preeclampsia by adenosine stress Magnetic Resonance Imaging and non-invasive methods like retinal vessel analysis, skin measurement of advanced glycation end products, flow-mediated dilation or pulse wave analysis in comparison to women after healthy pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 18-60 years
* 5-15 years postpartum

Exclusion Criteria:

* Atrioventricular block, chronic obstructive pulmonary disease, bronchial asthma
* Pregnancy and/or active breastfeeding
* Glaucoma disease, epilepsy
* In addition for MRI: metal implants, electric devices, intolerance of contrast media, claustrophobia, renal or hepatic dysfunction (GFR < 30 ml/min)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Woman 5-15 years after pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Myocardial perfusion | Day 2
  Measured by adenosine stress Magnetic Resonance Imaging (ml/min/g)

SECONDARY OUTCOMES:
Cardiac fibrosis | Day 2
  Measured by Magnetic Resonance Imaging (g)
Immune cell phenotypes | Day 1
  Measured in isolated peripheral blood mononuclear cells
Concentration of N-terminal prohormone of brain natriuretic peptide | Day 1
  Measured in serum (ng/l)
Concentration of brain natriuretic peptide | Day 1
  Measured in serum (ng/l)
Urinary protein | Day 1
  Measured in spot urine (mg)
Advanced glycation end products | Day 1
  Measured by skin autofluorescence (arbitrary units)
Body fat mass | Day 1
  Measured by bioimpedance analysis (%)
Body fat-free mass | Day 1
  Measured by bioimpedance analysis (%)
Hand grip strength | Day 1
  Measured by dynamometer (kg)
Systolic blood pressure | Day 1
  Mean of three consecutive blood pressure measurements (mmHg)
Diastolic blood pressure | Day 1
  Mean of three consecutive blood pressure measurements (mmHg)
Pulse wave velocity | Day 1
  Calculated by algorithm based on age and blood pressure values (m/s)
Flow-mediated dilation | Day 1
  Measured by brachial artery diameter (µm)
Reactive hyperemia index | Day 1
  Measured by finger plethysmography
Choroidal thickness | Day 1
  Measured with Optical Coherence Tomography (µm)
Macular volume | Day 1
  Measured with Optical Coherence Tomography (mm³)
Arterial dilation induced by retinal flicker stimulation | Day 1
  Measured with Dynamic Vessel Analyser (seconds)
Venous dilation induced by retinal flicker stimulation | Day 1
  Measured with Dynamic Vessel Analyser (seconds)

CONTACTS AND LOCATIONS:
Overall Officials: Anja Mähler, PhD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Experimental and Clinical Research Center, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of reported articles (text, tables, figures, supplemental data) will be shared after deidentification.
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.